CLINICAL TRIAL: NCT02633033
Title: A Prospective Observational Registry of H.P. Acthar® Gel for the Treatment of Multiple Sclerosis Relapse
Brief Title: Observational Registry of Acthar Gel for Participants With Multiple Sclerosis Relapse
Status: Completed | Type: Observational
Sponsor: Mallinckrodt (Industry)
Collaborators: Mallinckrodt ARD Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: MNK14130050
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; Relapsing-Remitting; Acthar; Corticotropin; MS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Acthar Gel was first approved by the Food and Drug Administration in 1952.

It has been used to treat many different illnesses, including multiple sclerosis.

This study will observe how treatment with Acthar affected the daily lives of patients who suffer with relapsing/remitting MS.

It will collect information on symptoms, recovery, treatment patterns and safety outcomes.

DETAILED DESCRIPTION:
Acthar Gel (repository corticotropin injection) contains a non-bovine analogue of adrenocorticotropic hormone (ACTH) for intramuscular or subcutaneous use.

It was initially approved by the FDA in 1952 and is used for multiple indications.

This registry will evaluate the use of Acthar Gel for the treatment of MS exacerbations in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female ≥ 18 years of age.
2. Patient has a clinically definite relapsing form of Multiple Sclerosis according to McDonald Criteria (2010 revision).
3. Patient with an acute MS exacerbation as determined by their treating clinician.
4. Patient planning to initiate Acthar Gel for the treatment of an acute MS exacerbation.
5. Patient capable of providing informed consent.

Exclusion Criteria:

1. Patients with a diagnosis of Progressive MS.
2. Patients that require concomitant corticosteroid therapy.
3. Patients receiving experimental drug therapy.
4. Patients with a history of scleroderma, systemic fungal infections, ocular herpes simplex within prior 5 years.
5. Patient has any solid tumor malignancy currently diagnosed or undergoing therapy, or has received therapy for any solid tumor malignancy in the 5 years prior to the Enrollment Visit, with the exception of treated and cured basal cell carcinoma, treated and cured squamous cell carcinoma of the skin, and treated and cured carcinoma in situ of the cervix.
6. Patients who had recent surgery or have a history of or the presence of a peptic ulcer within 6 months prior to study entry, congestive heart failure, or sensitivity to proteins of porcine origin.
7. If female, pregnant or breast-feeding; or, if of childbearing age, an unwillingness to use appropriate birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a relapsing form of MS who initiate treatment with Acthar Gel for an MS exacerbation
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-05-09 (Actual)

PRIMARY OUTCOMES:
Physical subscale score of the Multiple Sclerosis Impact Scale, v.1 (MSIS-29v1) | at 2 months
  Participants rate 20 physical symptoms of multiple sclerosis (MS) on a scale from 1=not at all to 5=extremely. The highest possible score is 100. Higher scores mean physical symptoms of MS have a higher impact on day-to-day life.
  For patients having a relapse during the study period, the schedule of assessments restarts at the time of relapse(s).

SECONDARY OUTCOMES:
Physical subscale score of the MSIS-29v1 within 6 months | within 6 months
  Participants rate 20 physical symptoms of MS on a scale from 1=not at all to 5=extremely. The highest possible score is 100. Higher scores mean physical symptoms of MS have a higher impact on day-to-day life.
  For patients having a relapse during the study period, the schedule of assessments restarts at the time of relapse(s).
  Rows: at 2 weeks, at 1 Month, at 3 Months, at 4 Months, at 5 Months, at 6 Months
Psychological subscale score of the MSIS-29v1 within 6 months | within 6 months
  Participants rate 9 psychological symptoms of MS on a scale from 1=not at all to 5=extremely. The highest possible score is 45. Higher scores mean psychological symptoms of MS have a higher impact on day-to-day life.
  For patients having a relapse during the study period, the schedule of assessments restarts at the time of relapse(s).
  Rows: at 2 weeks, at 1 Month, at 2 months, at 3 Months, at 4 Months, at 5 Months, at 6 Months
Score on the Expanded Disability Status Scale/Functional System Score (EDSS/FSS) | within 6 months
  Treating clinicians trained in completing the EDSS/FSS (neurologist or other healthcare professional such as a nurse practitioner or physician assistant) complete the EDSS/FSS to evaluate patient neurologic impairment.
  The EDSS is based on the standard neurological examination and is used by the clinician in conjunction with the Functional System Score (FSS) to produce a disability score. The FSS is a companion scale that is part of the EDSS
  Expanded Disability Status Scale (EDSS) is a well validated 10 point ordinal clinical rating scale with scores ranging from 0 (normal neurological examination) to 10 (death due to MS) in 0.5 point increments. The highest possible score is 100. A higher score means more neurological disability.
  For patients having a relapse during the study period, the schedule of assessments restarts at the time of relapse(s).
  Rows: at Baseline, at 2 Months, at 6 Months
Clinical Global Impression of Improvement Scale (CGI-I) | within 6 months
  Treating clinicians complete the CGI-I. It is a scale that compares the overall condition of the patient to baseline. Scores range from 1 (very much improved) to 7 (very much worse). The highest possible score is 7. Lower scores mean improvement.
  For patients having a relapse during the study period, the schedule of assessments restarts at the time of relapse(s).
  Rows: at Baseline, at 2 Months, at 6 Months
Total score of the MSIS-29v1 within 6 months | within 6 months
  Participants rate 29 psychological symptoms of MS on a scale from 1=not at all to 5=extremely. The highest possible score is 145. Higher scores mean total symptoms of MS have a higher impact on day-to-day life.
  For patients having a relapse during the study period, the schedule of assessments restarts at the time of relapse(s).
  Rows: at 2 weeks, at 1 Month, at 2 months, at 3 Months, at 4 Months, at 5 Months, at 6 Months
Number of participants with treatment response based on the MSIS-29v1 physical subscale score | within 6 months
  Treatment response is defined as an 8-point improvement on the MSIS-29v1 physical subscale score at 2 weeks and 1, 2, 3, 4, 5 and 6 months.
  For patients having a relapse during the study period, the schedule of assessments restarts at the time of relapse(s).
Number of participants with treatment response based on the EDSS | within 6 months
  Treatment response is defined as a 0.5 point improvement on the EDSS at 2 and 6 months.
  For patients having a relapse during the study period, the schedule of assessments restarts at the time of relapse(s).
  Rows: at 2 Months, at 6 Months
Percent of normal work hours missed (absenteeism) due to MS exacerbation | within 6 months
  For patients having a relapse during the study period, the schedule of assessments restarts at the time of relapse(s).
  Rows: at 2 weeks, at 1 Month, at 2 Months, at 3 Months, at 4 Months, at 5 Months, at 6 Months
Number of participants with impairment at work and/or reduced on-the-job effectiveness (presenteeism) due to MS exacerbation | within 6 months
  For patients having a relapse during the study period, the schedule of assessments restarts at the time of relapse(s).
  Rows: at 1 Week, at 2 Weeks, at 3 Weeks, at 4 Weeks, at 6 Weeks, at 2 Months, at 3 Months, at 4 Months, at 5 Months, at 6 Months
Number of participants with overall Impairment at Work (absenteeism + presenteeism) due to MS exacerbation | within 6 months
  For patients having a relapse during the study period, the schedule of assessments restarts at the time of relapse(s).
  Rows: at 1 Week, at 2 Weeks, at 3 Weeks, at 4 Weeks, at 6 Weeks, at 2 Months, at 3 Months, at 4 Months, at 5 Months, at 6 Months
Number of participants with Impairment in activities other than work due to MS exacerbation | within 6 months
  For patients having a relapse during the study period, the schedule of assessments restarts at the time of relapse(s).
  Rows: at 1 Week, at 2 Weeks, at 3 Weeks, at 4 Weeks, at 6 Weeks, at 2 Months, at 3 Months, at 4 Months, at 5 Months, at 6 Months
Number of days per month an unpaid caregiver missed work due to the patient's MS | within 6 months
  For patients having a relapse during the study period, the schedule of assessments restarts at the time of relapse(s).
Number of MS-related off-site clinical/office visits with a specialist or a general practitioner | within 6 months
  For patients having a relapse during the study period, the schedule of assessments restarts at the time of relapse(s).
Number of MS-related healthcare professional visits at home | within 6 months
  For patients having a relapse during the study period, the schedule of assessments restarts at the time of relapse(s).
Number of MS-related emergency department visits | within 6 months
  For patients having a relapse during the study period, the schedule of assessments restarts at the time of relapse(s).
Number of MS-related hospitalizations | within 6 months
  For patients having a relapse during the study period, the schedule of assessments restarts at the time of relapse(s).
Number of MS-related MRIs | within 6 months
  For patients having a relapse during the study period, the schedule of assessments restarts at the time of relapse(s).
Number of days per month of MS-related paid and unpaid caregiver assistance | within 6 months
  For patients having a relapse during the study period, the schedule of assessments restarts at the time of relapse(s).

CONTACTS AND LOCATIONS:
Overall Officials: Study Directo, Study Director — Mallinckrodt
Locations (38):
- United States (38):
  - Alabama Neurology Associates, Homewood, Alabama
  - Territory Neurology & Research Institute, Tucson, Arizona
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - Advanced Neurosciences Research, Fort Collins, Colorado
  - Associated Neurologists of Southern Connecticut, Fairfield, Connecticut
  - MedStar Health, Washington D.C., District of Columbia
  - Emery Neuroscience Center, Lighthouse PT, Florida
  - Neurology Associates, Maitland, Florida
  - Cordova Research Institute, Miami, Florida
  - Collier Neurologic Specialists, Naples, Florida
  - Florida Neurological Center, Ocala, Florida
  - Neurological Services of Orlando, Orlando, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Negroski, Sutherland and Hanes Neurology, Sarasota, Florida
  - Infinity Clinical Research, Sunrise, Florida
  - Columbus Research & Wellness Institute, Columbus, Georgia
  - Neurology of Central Georgia, Macon, Georgia
  - Meridian Clinical Research, Savannah, Georgia
  - College Park Family Care Center, Overland Park, Kansas
  - University System of Maryland, Baltimore, Maryland
  - International Neurorehabilitation Institute, Lutherville, Maryland
  - Neurology Center of New England, Foxborough, Massachusetts
  - Milford Regional Medical Center, Hopedale, Massachusetts
  - Detroit Clinical Research Center, Farmington Hills, Michigan
  - CentraState Medical Center, Freehold, New Jersey
  - Strotira, Inc., New York, New York
  - Alpha Neurology, Staten Island, New York
  - Five Towns Neurology, Woodmere, New York
  - Braunstein Neurology, Mooresville, North Carolina
  - The Toledo Clinic, Toledo, Ohio
  - Oak Clinic for Multiple Sclerosis, Uniontown, Ohio
  - Optimum Neurology, Bala-Cynwyd, Pennsylvania
  - Irene Greenhouse MD, Jamison, Pennsylvania
  - Neurology and Stroke Associates, Lititz, Pennsylvania
  - D. Gary Kolva, MD, Neurology, West Reading, Pennsylvania
  - Colonial Healthcare, Sumter, South Carolina
  - Ogden Clinic, Ogden, Utah
  - Dominion Neurological Services, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaplan J, Miller T, Baker M, Due B, Zhao E. Repository corticotropin injection improves quality metrics in an observational study of multiple sclerosis relapse. Neurodegener Dis Manag. 2021 Dec;11(6):469-476. doi: 10.2217/nmt-2021-0030. Epub 2021 Dec 3. PMID 34860120
- [Derived] Kaplan J, Miller T, Baker M, Due B, Zhao E. A Prospective Observational Registry of Repository Corticotropin Injection (Acthar(R) Gel) for the Treatment of Multiple Sclerosis Relapse. Front Neurol. 2020 Dec 22;11:598496. doi: 10.3389/fneur.2020.598496. eCollection 2020. PMID 33414758